CLINICAL TRIAL: NCT06591598
Title: An Open-label, Non-randomized, Multi-center, Phase 4 Pharmacokinetic Study to Evaluate the Systemic Exposure After Bilateral Intravitreal Administration of High Dose (8 mg) Aflibercept in Adults With Diabetic Macular Edema or Neovascular Age-related Macular Degeneration
Brief Title: A Study to Learn About the Blood Levels of Aflibercept When High-dose Aflibercept is Injected in Both Eyes of Participants With Diabetic Macular Edema or Neovascular Age-related Macular Degeneration
Acronym: DEUTERON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22578; 2024-511665-11-00 (Registry Identifier: CTIS(EU))
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Macular Edema; Neovascular Age-related Macular Degeneration
Keywords: Diabetic macular edema (DME); Neovascular age-related macular degeneration (nAMD)
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen 1 (Experimental): 15 participants will be assigned to Regimen 1. Regimen 1 participants will be administered 8 mg aflibercept injections according to the Regimen 1 dosing schedule.
  Interventions: Drug: Aflibercept (BAY86-5321, Eylea)
- Regimen 2 (Experimental): Up to 15 participants will be assigned to Regimen 2. Regimen 2 participants will be administered 8 mg aflibercept injections according to the Regimen 2 dosing schedule.
  Interventions: Drug: Aflibercept (BAY86-5321, Eylea)
- Regimen 3 (Experimental): Up to 15 participants will be assigned to Regimen 3. Regimen 3 participants will be administered 8 mg aflibercept injections according to the Regimen 3 dosing schedule.
  Interventions: Drug: Aflibercept (BAY86-5321, Eylea)

INTERVENTIONS:
Drug: Aflibercept (BAY86-5321, Eylea) — 8 mg, intravitreal injection
  Other Names: BAY86-5321, Eylea HD

SUMMARY:
Researchers are looking for a better way to treat participants who have diabetic macular edema (DME) or neovascular age-related macular degeneration (nAMD).

DME is a diabetes-related eye disorder. In DME, the macula swells up due to fluid leakage from damaged blood vessels, resulting in vision problems. DME is a leading cause of vision loss in working age adults. nAMD is an eye disorder that causes vision loss due to the growth of abnormal blood vessels that leak blood or retinal fluid into the macula (the central part of the retina). nAMD is a leading cause of vision loss for people aged 50 and older.

The study treatment Aflibercept (also called BAY 86-5321) is a drug that blocks a protein called vascular endothelial growth factor (VEGF) which causes abnormal growth and leakage of blood vessels at the back of the eye.

The main purpose of this study is to to collect more information on the blood levels of aflibercept when 8 mg aflibercept is injected in both eyes of participants with DME or nAMD.

For this, the researchers will analyze Maximum observed concentration (Cmax): the highest amount of aflibercept in participants' blood will be measured after multiple doses of aflibercept during the study.

Participants will receive 8 mg aflibercept as injections into the vitreous cavity (jelly-like substance that fills the centre of the eye) of both eyes.

Participants will be divided into three groups and will receive initial and maintenance injections of 8 mg aflibercept in both eyes. Researchers will closely monitor the health of the participants during the study.

During the study, the doctors and their study team will:

* take blood and urine samples
* do physical examinations
* examine heart health using electrocardiogram (ECG)
* check vital signs such as blood pressure, heart rate, body temperature
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years of age (or country's legal age of adulthood if the legal age is >18 years).
* Participants (treatment naïve or previously treated) requiring intravitreal anti-vascular endothelial growth factor (VEGF) treatment in both eyes in the opinion of the investigator.
* Participants with type 1 or type 2 diabetes mellitus and DME in both eyes with active central involvement (CI-DME) in at least one eye with central retinal thickness (CRT) ≥300 µm (or ≥320 µm on Spectralis) as determined by the investigator at the screening visit, OR diagnosis of nAMD in both eyes with active subfoveal choroidal neovascularization (CNV) in at least one eye with intraretinal fluid (IRF) and/or subretinal fluid (SRF) on OCT as determined by the investigator at the screening visit.
* Best corrected visual acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) letter score of 78 to 24 (approximate Snellen equivalent of 20/32 to 20/320) in eyes with active disease and decreased vision determined to be primarily the result of DME or nAMD.
* A female participant is eligible to participate if she is not pregnant or breastfeeding. Women of childbearing potential (WOCBP) or men who are sexually active with partners of childbearing potential must agree to use highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 4 months after the last administration of study intervention.

Exclusion Criteria:

* Evidence of macular edema due to any cause other than diabetes mellitus in patients with DME or neovascular age-related macular degeneration in patients with nAMD in either eye.
* Active proliferative diabetic retinopathy (DR) in either eye.
* Panretinal laser photocoagulation (PRP) or macular laser photocoagulation in either eye with CI-DME or active nAMD within 12 weeks (84 days) of the screening visit.
* Prior treatment with intravitreal (IVT) 2 mg aflibercept (EYLEA) in either eye within 12 weeks (84 days) of the screening visit or with IVT 8 mg or HD aflibercept in either eye within 24 weeks (168 days) of the screening visit.
* Prior treatment with any other approved IVT agent with anti-VEGF effect (e.g. ranibizumab, bevacizumab, brolucizumab, faricimab, pegaptanib sodium or biosimilars) in either eye within 4 weeks (28 days) of the screening visit.
* Prior treatment with any ocular gene or cell therapy treatment in either eye.
* Previous use of intraocular or periocular corticosteroids in either eye within 16 weeks (112 days) of the screening visit, or OZURDEX® implant within 180 days of the screening visit or ILUVIEN® or RETISERT® implant at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of free aflibercept | Up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- Czechia (2):
  - Fakultní nemocnice Královské Vinohrady - Urologická klinikay, Prague
  - Axon Clinical, s.r.o., Prague
- Hungary (2):
  - Budapest Retina Associates, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Slovakia (2):
  - Univerzitna nemocnica Bratislava, Nem. Sv. Cyrila a Metoda, Bratislava
  - Fakultna nemocnica s poliklinikou Zilina, Žilina

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22578